CLINICAL TRIAL: NCT05386004
Title: Effects Of Focus On Birth-Specific Stereogram Cards (BSSC) On Perception Of Labour Pain
Brief Title: Labour Pain and Birth-Specific Stereogram Cards (BSSC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Esra Yurtsev, Asistant Professor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: interventional
Record Dates: First submitted 2022-04-14; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Labor Pain; Birth, First
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Two groups of primiparous pregnant women who met the inclusion criteria and agreed to participate in the study were included in the study. Pregnant women were randomly assigned to experimental and control groups. The experimental group was treated with BSSC.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BSSC group (Experimental): Participants in the experimental group were allowed to focus with BSSC during uterine contractions in the first stage of labor.
  Interventions: Other: Birth-Specific Stereogram Cards (BSSC)
- control group (No Intervention): The participants in the control group were provided with routine care in the first stage of labor. No intervention was made.

INTERVENTIONS:
Other: Birth-Specific Stereogram Cards (BSSC) — Focus on Birth-Specific Stereogram Cards (BSSC) during uterine contractions in latent active and transitional phase
  Arms: BSSC group

SUMMARY:
Background: Reducing the perception of labour pain is important to reduce the negative consequences of labour pain and to increase women's satisfaction with the birth experience. Two-dimensional (2D) images (Stereogram) that create the three-dimensional (3D) perception in the mind may be effective in reducing the perception of labour pain.

Objectives: This study is conducted for purpose of determining the effect of focus on the birth-specific stereogram cards (BSSC), on perception of labour pain.

Methods: This research is an experimental prospective randomized controlled clinical study. The research was conducted at the delivery room of a state hospital in Istanbul. Pregnant women, who agreed to participate in the study and met the study criteria, were included in the study, as 30 ones were in the experimental group (BSSC group) and 30 ones were in the control group. The Pregnancy Data Form, State Anxiety Scale, BSSC, • PRS Review Comments Visual Analog Scale(VAS), Postpartum Data Form were used as data collection tools. The BSSC in birth are designed by researchers and are created using the stereogram creator program. BSSC's 10 cards set with different patterns and silhouettes on the background. The analyses were performed, using SPSS software version 20.

KEY WORDS: Birth, Labour pain, Birth-specific stereogram cards, Stereogram card, Focus on birth.

DETAILED DESCRIPTION:
Introduction Labour pain is not only sensory, but a multifaceted subjective phenomenon having emotional, motivational and cognitive dimensions .The American Academy of Obstetrics and Gynecology (ACOG) and the Society of Anesthesiology (ASA) report that labour pain should be remedied by a therapy due to the maternal and fetal effects of the severe labour pain. In the management of labour pain, non-pharmacological approaches are aiming to increase maternal satisfaction, control feeling in birth and sufficiency sense, and to reduce obstetric interventions. Distraction and cognitive strategies are used to prevent the transmission of painful stimuli information to the central nervous system. In painful situations, pain transmission is prevented by distracting the attention from pain ensuring focus stimuli other pain in transmission by focusing on stimuli outside the pain.

Distraction during delivery includes the process of removing a woman's attention from the pain of birth by means of any external stimuli. Especially, determination of a focal spot enables to maintain the concentration. Images can be the focus of any object. It is seen that the "plippets" cards known as the "distraction cards" and virtual realityare used in reducing the perceived pain level. However, there was no study showing the effect of "focus and distraction" on the perceived labour pain. The stereoscopic vision technique discovered by Charles Wheatstone in 1838 is also based on focus. Stereogram is the general name of two-dimensional (2D) images that create three-dimensional (3D) perception in the mind. A person can focus the lenses on the stereograms of the lenses, zoom the eyeballs to a distant point located behind the stereogram image and thus trick the brain and allow the brain view the 3D images.The stereograms known as "squint at and be surprised" in Turkey in the 90s were popular in the "magic eye" series especially in the USA .

There are different methods to view the targeted three-dimensional image in the stereogram. Some people may see the images simply in a stereogram, while others have to educate their eyes to separate the eye convergence resulting from the focus of the lens. One of the methods that may be used is to hold the image against face so that the nose contacts with the image. Most people cannot focus on the image, while the image is too close to their eyes. If the person moves the image away from his/her face slowly, the brain will focus on pairs of patterns that correspond to the degree of convergence of the two eyeballs at one point. Another method is to look constantly at an object behind the image to obtain the suitable degree of convergence while keeping the field of view constant on the image for purpose of convincing the brain to focus on the image. In a modified method, the person constantly looks at his/her own reflection on the bright surface. Thus, it shall be ensured that the brain achieves the necessary degree of convergence when focus on the near field, and that the three-dimensional image behind the pattern is visible.

On the basis of the stereoscopic vision technique, it is thought that focusing on the stereogram cards specially prepared for birth can also be effective in reducing the labour pain perception. In this study, researchers aim to determine the effect of focusing on birth-specific stereogram cards(BSSC) on labour pain perception.

Methods Study design This research is an experimental prospective randomized controlled clinical study.

Sample and Setting The research was conducted at the delivery room of a state hospital in Istanbul. In the delivery room where the work was conducted, 528 nulliparous women gave the vaginal birth. At the time of the research the standard midwifery care provided in the hospital during birth.

60 pregnant women, who agreed to participate in the study and met the study criteria, were included in the study, as 30 ones were in the test group (BSSC group) and 30 ones were in the control group. Power analysis is performed in the PASS program to determine the number of samples of the study.

According to previous studies, it is assumed that the difference between the level of pain between the experimental (BSSC) group and the control group is 5 after the intervention and the standard deviation of the control and the experimental group at the first measurement is 2. It is determined that, when the significance level α = 0.05 is taken as the power of 1-β = 0.99, the sample size is 30 for the control group and 30 for the experimental group. The research findings are limited to the research sample, can not be generalized.

İnterventions The pregnant women, who agreed the study, were included in randomization. All applicant is given a barcode number in the polyclinic. This barcode number was used for randomization. Single numbers were included in the experimental group, double in the numbers control group. The participants in the BSSC group were given a practical training on the focus technique on stereogram cards for one hour in the prenatal final trimester. The participants in the BSSC group were admitted to the delivery room when the birth process started. It was ensured that the participants in the BSSC group were focus on contractions in the latent phase, active phase and the transition phase by BSSC throughout. The participants in the BSSC group were admitted a pain assessment via VAS every two hours before and after the focus in parallel with clinical routine practice. A VAS was administered to the delivery room in the first admission and every two hours after birth without any interference to the participant in the control group. The state anxiety scale was assessed to both groups when cervical dilatation was 3-4 cm in the latent phase and cervical dilatation was 8-9 cm in the transition phase. Postpartum fatigue level and satisfaction of participants from birth were applied to both groups at the 2nd hour postpartum.

Data Collection The Pregnancy Data Form, State Anxiety Scale, BSSC, VAS, Postpartum Data Form were used as data collection tools.

The Pregnancy Data Form was prepared based on the literature. It consists of questions about the socio-demographic characteristics, medical and obstetric characteristics of the pregnant wo man, information and thoughts about the current pregnancy and birth.

Intrapartum Process Data Form includes about Gestational week, date and time of birth pain, drugs and applications in the first stage of labour, table before and after the application of stereogram card (cervical dilatation and wiping, level of head and condition of membranes, severity and frequency of contractions, fetal heart rate ( FKA), the mother's vital signs and behaviors during labour), the time when the second stage begins, the end time, the total duration of labour.

State Anxiety Scale was used to measure the level of anxiety experienced by pregnant women in both groups in the first stage of labour. According to the severity of the individual's emotions or behaviors in the situation he / she is experiencing, (1) None, (2) Some, (3) Many and (4) Completely requires to answer by marking one of the options. The state anxiety scale consists of 20 statements. The score obtained from the scale can vary between 20 and 80. The larger the score, the higher the anxiety level, the smaller the lower the level of anxiety.

VAS is a scale used to measure perceived pain. It was used in the studies to evaluate the perceived birth pain. It was found to be valid and reliable. In the form of a 0-10cm ruler, one end of the scale indicates 0 painlessness and the other 10 indicates the most severe degree of pain intensity.

Postpartum evaluation data form was prepared to evaluate the birth process for the participants of BSSC group and control group. At the end of the 2nd hour, the pregnant woman's thoughts about this birth, her thoughts about the labour pain, how she felt at the end of the birth and her satisfaction with the practices performed during the labour are included.

Design of BSSC The structure of the stereograms consists of two images. One of them is a depth map and the other is a texture map. These two visual elements are combined with specially designed computer software. Birth-specific stereogram cards (BSSC) in birth are designed by researchers and are created using the stereogram creator program. In the BSSC design, it was used as a tissue image to attract the attention of the mothers, and the pregnant, father, baby silhouettes were used as oxytocic pictures. These three-dimensional visual images were revised and finalized in the pilot study. BSSC is designed as a set with images to facilitate the use of the mothers. BSSC's 10 cards set with different patterns and silhouettes on the background.

Ethical Considerations Pregnant Women have given their written informed consent. The study protocol has been approved by the ethical committee of the Şişli Hamidiye Etfal Education and Research Hospital, Study No: 569 on the 27th October 2015.

Data Analysis The analysis were performed, using SPSS software version 20 (Statistical Package for Social Sciences Inc, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

Pregnancy in term (37-42W)

* Have a fetus in a single, live and vertex position
* Latent stage of labour
* Cervical dilatation less than 5 cm
* Vaginal delivery planning
* No pregnancy complications
* Contractions have started and are regular
* No language problem
* Verbal communication
* Pregnant women accepted to study.

Exclusion Criteria:

Narcotic analgesic or sedative area

* Systemic disease such as heart disease, hypertension, diabetes, kidney disease
* Pregnant women with pregnancy complications (plascenta previa, preeclampsia, oligohydroamnios, polyhydroamnios, position / presentation disorder, etc.).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women who have started labor
Enrollment: 60 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Durations of stage of labour in Birth- Specific Stereogram Cards (BSSC) group and control group | during the first stage of birth (up to 12 hours)
  Comparison of latent, active and transitional phase times for the control and intervention groups. Measuring the effect of BSSC in shortening the birth time. It is desirable that the birth durations (latent, active and transitional phase) of the participants in the intervention group were short and meaningful for study
Comparison of Visual Analog Scale (VAS) score averages of the Birth- Specific Stereogram Cards (BSSC) group and control group | every two hours during the first stage of labor (during the first stage of birth (up to 12 hours)
  Comparison of VAS scores applied every two hours to the BSSC group and control groups during the latent active and transitional phases in the first stage of labour.
  VAS is a scale used to measure perceived pain. It was used in the studies to evaluate the perceived birth pain. It was found to be valid and reliable. In the form of a 0-10cm ruler, one end of the scale indicates 0 painlessness and the other 10 indicates the most severe degree of pain intensity.
Comparison of state anxiety and postpartum fatigue levels of the Birth- Specific Stereogram Cards(BSSC) group and control group | in the latent phases (an average of 1 hour after birth) transitional phases (an average of 9 hour after birth) in the first stage of labor.
  Comparison of The State Anxiety Scale scores applied to the Birth- Specific Stereogram Cards (BSSC) group and control groups in the latent and transitional phases in the first stage of labour.
  A high state anxiety scale score indicates a high level of anxiety, and a low score indicates a low level of anxiety.
  State Anxiety Scale was used to measure the level of anxiety experienced by pregnant women in both groups in the first stage of labour. According to the severity of the individual's emotions or behaviors in the situation he / she is experiencing, (1) None, (2) Some, (3) Many and (4) Completely requires to answer by marking one of the options. The state anxiety scale consists of 20 statements. The score obtained from the scale can vary between 20 and 80. The larger the score, the higher the anxiety level, the smaller the lower the level of anxiety.

SECONDARY OUTCOMES:
Evaluation of the opinions of the BSSC group participants about the BSSC application | 2 hours after birth (up to 2 hours)
  Application of a questionnaire consisting of questions measuring BSSC group participants' satisfaction with the BSSC application, whether they find the application effective, and whether they want to use BSSC in their next birth.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Atlas University, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All data on the study will be published and shared in a journal.

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists Committee on Obstetric Practice. ACOG committee opinion. No. 339: Analgesia and cesarean delivery rates. Obstet Gynecol. 2006 Jun;107(6):1487-8. doi: 10.1097/00006250-200606000-00060. PMID 16738188
- [Background] Alp, N., Mete, S. (2008). Effect of Postpartum Fatigue Level, Sleep and Nutrition on Fatigue. The Journalof the Nursing School, Ataturk University, 11(4).
- [Background] Altunoglu, S. (2017) Stereogram types and structures. Access: 10.01.2017. https://www.academia.edu/16704677/
- [Background] ASA. (2010). American Society of Anesthesia. Committee of Origin: Obstetrical Anesthesia (Approved by the ASA House of Delegates on October 13, 1999 and last amended on October 20. 2010.
- [Background] Beevi Z, Low WY, Hassan J. The Effectiveness of Hypnosis Intervention for Labor: An Experimental Study. Am J Clin Hypn. 2017 Oct;60(2):172-191. doi: 10.1080/00029157.2017.1280659. PMID 28891771
- [Background] Boaviagem A, Melo Junior E, Lubambo L, Sousa P, Aragao C, Albuquerque S, Lemos A. The effectiveness of breathing patterns to control maternal anxiety during the first period of labor: A randomized controlled clinical trial. Complement Ther Clin Pract. 2017 Feb;26:30-35. doi: 10.1016/j.ctcp.2016.11.004. Epub 2016 Nov 11. PMID 28107846
- [Background] Canbulat N, Inal S, Sonmezer H. Efficacy of distraction methods on procedural pain and anxiety by applying distraction cards and kaleidoscope in children. Asian Nurs Res (Korean Soc Nurs Sci). 2014 Mar;8(1):23-8. doi: 10.1016/j.anr.2013.12.001. Epub 2013 Dec 14. PMID 25030489
- [Background] Chaillet N, Belaid L, Crochetiere C, Roy L, Gagne GP, Moutquin JM, Rossignol M, Dugas M, Wassef M, Bonapace J. Nonpharmacologic approaches for pain management during labor compared with usual care: a meta-analysis. Birth. 2014 Jun;41(2):122-37. doi: 10.1111/birt.12103. Epub 2014 Apr 25. PMID 24761801
- [Background] Choudhury N, Amer I, Daniels M, Wareing MJ. Audiovisual distraction reduces pain perception during aural microsuction. Ann R Coll Surg Engl. 2013 Jan;95(1):34-6. doi: 10.1308/003588413X13511609955535. PMID 23317724
- [Background] Creehan, P.A. (2007). Pain Relief and Comfort Measure in Labour. In: Kathleen Rice Simpson, Patricia A. Creehan (3rd Ed).Awhonn's Perinatal Nursing;: 333-460p.
- [Background] Fahami F, Behmanesh F, Valiani M, Ashouri E. Effect of heat therapy on pain severity in primigravida women. Iran J Nurs Midwifery Res. 2011 Winter;16(1):113-6. PMID 22039388
- [Background] Finlayson K, Downe S, Hinder S, Carr H, Spiby H, Whorwell P. Unexpected consequences: women's experiences of a self-hypnosis intervention to help with pain relief during labour. BMC Pregnancy Childbirth. 2015 Sep 25;15:229. doi: 10.1186/s12884-015-0659-0. PMID 26407981
- [Background] Floris L, Irion O, Courvoisier D. Influence of obstetrical events on satisfaction and anxiety during childbirth: a prospective longitudinal study. Psychol Health Med. 2017 Sep;22(8):969-977. doi: 10.1080/13548506.2016.1258480. Epub 2016 Nov 17. PMID 27855515
- [Background] Gantz L, Bedell HE. Transfer of perceptual learning of depth discrimination between local and global stereograms. Vision Res. 2010 Aug 23;50(18):1891-9. doi: 10.1016/j.visres.2010.06.011. Epub 2010 Jun 25. PMID 20600234
- [Background] Gomez AT, Lupon N, Cardona G, Aznar-Casanova JA. Visual mechanisms governing the perception of auto-stereograms. Clin Exp Optom. 2012 Mar;95(2):146-52. doi: 10.1111/j.1444-0938.2011.00664.x. Epub 2011 Oct 24. PMID 22023025
- [Background] Grossman, M., Smith, C. (2004). Magic Eye Beyond 3D: Improve Your Vision. Kansas City: Andrews Mc Meel Publishing; ISBN 0-7407-4527-1.
- [Background] Guo C, Deng H, Yang J. Effect of virtual reality distraction on pain among patients with hand injury undergoing dressing change. J Clin Nurs. 2015 Jan;24(1-2):115-20. doi: 10.1111/jocn.12626. Epub 2014 Jun 4. PMID 24899241
- [Background] Moghimi-Hanjani S, Mehdizadeh-Tourzani Z, Shoghi M. The Effect of Foot Reflexology on Anxiety, Pain, and Outcomes of the Labor in Primigravida Women. Acta Med Iran. 2015 Aug;53(8):507-11. PMID 26545996
- [Background] Jahdi F, Sheikhan F, Haghani H, Sharifi B, Ghaseminejad A, Khodarahmian M, Rouhana N. Yoga during pregnancy: The effects on labor pain and delivery outcomes (A randomized controlled trial). Complement Ther Clin Pract. 2017 May;27:1-4. doi: 10.1016/j.ctcp.2016.12.002. Epub 2016 Dec 23. PMID 28438273
- [Background] Karlstrom A, Nystedt A, Hildingsson I. A comparative study of the experience of childbirth between women who preferred and had a caesarean section and women who preferred and had a vaginal birth. Sex Reprod Healthc. 2011 Aug;2(3):93-9. doi: 10.1016/j.srhc.2011.03.002. Epub 2011 Apr 3. PMID 21742287
- [Background] Kheirkhah M, Vali Pour NS, Nisani L, Haghani H. Comparing the effects of aromatherapy with rose oils and warm foot bath on anxiety in the first stage of labor in nulliparous women. Iran Red Crescent Med J. 2014 Aug 17;16(9):e14455. doi: 10.5812/ircmj.14455. eCollection 2014 Sep. PMID 25593713
- [Background] Klomp T, Mannien J, de Jonge A, Hutton EK, Lagro-Janssen AL. What do midwives need to know about approaches of women towards labour pain management? A qualitative interview study into expectations of management of labour pain for pregnant women receiving midwife-led care in the Netherlands. Midwifery. 2014 Apr;30(4):432-8. doi: 10.1016/j.midw.2013.04.013. Epub 2013 Jun 19. PMID 23790961
- [Background] Koelewijn JM, Sluijs AM, Vrijkotte TGM. Possible relationship between general and pregnancy-related anxiety during the first half of pregnancy and the birth process: a prospective cohort study. BMJ Open. 2017 May 9;7(5):e013413. doi: 10.1136/bmjopen-2016-013413. PMID 28490549
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307
- [Background] Liossi, C., Franck, L.S. (2017). Psychological interventions for acute pediatric pain. Chapter 16.Access: 23. 07. 2017. http://cw.tandf.co.uk/clinicalpainmanagement/acute-pain/AcuteCh16.pdf.
- [Background] Long-Bellil L, Mitra M, Iezzoni LI, Smeltzer SC, Smith LD. Experiences and unmet needs of women with physical disabilities for pain relief during labor and delivery. Disabil Health J. 2017 Jul;10(3):440-444. doi: 10.1016/j.dhjo.2017.02.007. Epub 2017 Apr 6. PMID 28428112
- [Background] Lowe NK, Corwin EJ. Proposed biological linkages between obesity, stress, and inefficient uterine contractility during labor in humans. Med Hypotheses. 2011 May;76(5):755-60. doi: 10.1016/j.mehy.2011.02.018. Epub 2011 Mar 5. PMID 21382668
- [Background] McCauley M, Stewart C, Kebede B. A survey of healthcare providers' knowledge and attitudes regarding pain relief in labor for women in Ethiopia. BMC Pregnancy Childbirth. 2017 Feb 7;17(1):56. doi: 10.1186/s12884-017-1237-4. PMID 28173771
- [Background] Melzac, R., 1999. From the gate to the neuromatrix. Pain;1999:82, 121-126p. Metinoglu, M., Irmak, A.Y., Kaya, SA. (2017). Application of Non-Pharmacological Methods to Give Birth in a Nulliparous Pregnancy. ACU Health Science Journal; 3:173-184p.
- [Background] Moayedi M, Davis KD. Theories of pain: from specificity to gate control. J Neurophysiol. 2013 Jan;109(1):5-12. doi: 10.1152/jn.00457.2012. Epub 2012 Oct 3. PMID 23034364
- [Background] Moberg, U.K. (2003). The Oxytocin factor: Tapping The hormone of Calm, Love and healing. De capo press.
- [Background] Oliveira NC, Santos JL, Linhares MB. Audiovisual distraction for pain relief in paediatric inpatients: A crossover study. Eur J Pain. 2017 Jan;21(1):178-187. doi: 10.1002/ejp.915. Epub 2016 Jul 26. PMID 27461092
- [Background] Ravangard R, Basiri A, Sajjadnia Z, Shokrpour N. Comparison of the Effects of Using Physiological Methods and Accompanying a Doula in Deliveries on Nulliparous Women's Anxiety and Pain: A Case Study in Iran. Health Care Manag (Frederick). 2017 Oct/Dec;36(4):372-379. doi: 10.1097/HCM.0000000000000188. PMID 28961642
- [Background] Risaw L, Narang K, Thakur JS, Ghai S, Kaur S, Bharti B. Efficacy of Flippits to Reduce Pain in Children during Venipuncture - A Randomized Controlled Trial. Indian J Pediatr. 2017 Aug;84(8):597-600. doi: 10.1007/s12098-017-2335-z. Epub 2017 Apr 5. PMID 28378139
- [Background] Sahiner NC, Bal MD. The effects of three different distraction methods on pain and anxiety in children. J Child Health Care. 2016 Sep;20(3):277-85. doi: 10.1177/1367493515587062. Epub 2015 Jun 2. PMID 26040282
- [Background] Shahoei R, Shahghebi S, Rezaei M, Naqshbandi S. The effect of transcutaneous electrical nerve stimulation on the severity of labor pain among nulliparous women: A clinical trial. Complement Ther Clin Pract. 2017 Aug;28:176-180. doi: 10.1016/j.ctcp.2017.05.004. Epub 2017 May 18. PMID 28779926
- [Background] Shaw-Battista J. Systematic Review of Hydrotherapy Research: Does a Warm Bath in Labor Promote Normal Physiologic Childbirth? J Perinat Neonatal Nurs. 2017 Oct/Dec;31(4):303-316. doi: 10.1097/JPN.0000000000000260. PMID 28520654
- [Background] Shourab NJ, Zagami SE, Golmakhani N, Mazlom SR, Nahvi A, Pabarja F, Talebi M, Rizi SM. Virtual reality and anxiety in primiparous women during episiotomy repair. Iran J Nurs Midwifery Res. 2016 Sep-Oct;21(5):521-526. doi: 10.4103/1735-9066.193417. PMID 27904638
- [Background] Simpson, K.R., O'brien-Abel, N. (2014). Labour and Birth. Simpson KR, Creehan PA. (4th Ed.), AWHONN Perinatal Nursing ; 344-510p.
- [Background] Snelgrove-Clarke, E., Budin, W. (2015). Labour and Childbirth. In: Evans R.J, Evans M.K, Brown Y (2nd Ed.). Canadian Maternity Newborn&Women's Health Nursing: 379-618p.
- [Background] Tzeng YL, Yang YL, Kuo PC, Lin YC, Chen SL. Pain, Anxiety, and Fatigue During Labor: A Prospective, Repeated Measures Study. J Nurs Res. 2017 Feb;25(1):59-67. doi: 10.1097/jnr.0000000000000165. PMID 28072678
- [Background] Tzeng YL, Chao YM, Kuo SY, Teng YK. Childbirth-related fatigue trajectories during labour. J Adv Nurs. 2008 Aug;63(3):240-9. doi: 10.1111/j.1365-2648.2008.04732.x. PMID 18702771
- [Background] Unalmis Erdogan S, Yanikkerem E, Goker A. Effects of low back massage on perceived birth pain and satisfaction. Complement Ther Clin Pract. 2017 Aug;28:169-175. doi: 10.1016/j.ctcp.2017.05.016. Epub 2017 Jun 1. PMID 28779925
- [Background] Vaziri F, Shiravani M, Najib FS, Pourahmad S, Salehi A, Yazdanpanahi Z. Effect of Lavender Oil Aroma in the Early Hours of Postpartum Period on Maternal Pains, Fatigue, and Mood: A Randomized Clinical Trial. Int J Prev Med. 2017 May 4;8:29. doi: 10.4103/ijpvm.IJPVM_137_16. eCollection 2017. PMID 28567231
- [Background] Webber AL, Wood J. Amblyopia: prevalence, natural history, functional effects and treatment. Clin Exp Optom. 2005 Nov;88(6):365-75. doi: 10.1111/j.1444-0938.2005.tb05102.x. PMID 16329744
- [Background] Zauderer, C.R. (2016). maximizing Comfort for the labouring woman. In: Lowdermilk, LD., Perry, ES., Cashion, K., Alden, KR. Maternity women's health care. 11. edition; 381-454p.